CLINICAL TRIAL: NCT05026931
Title: Effects of Foam Rolling Versus Stretching Exercises on Quadriceps, Hamstrings and Calf Muscle Length in University Sport's Students
Brief Title: Effects of Foam Rolling Versus Stretching Exercises on Quadriceps, Hamstrings and Calf Muscle Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/0407 Nubara
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Muscle Tightness
Keywords: Foam rolling Stretching exercises Calf Muscle length
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Foam Rolling
  Interventions: Other: Foam rolling
- Group B (Active Comparator): Stretching exercises
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Foam rolling — Group A will be treated with foam rolling effect on quadriceps, hamstring and calf muscle length. 5 min cycle ergometry, 6 min foam rolling 3 times for 30sec.For three session per week will be given atleast for 2 months.
  Arms: Group A
Other: Stretching exercises — Group B will be treated with stretching exercises effect on quadriceps, hamstring and calf muscle length. 5 min cycle ergometry, 6 min foam rolling 3 times for 30sec.For three session per week will be given atleast for 2 months.
  Arms: Group B

SUMMARY:
This project will be Randomized control trial conducted to check the effects of foam rolling and stretching exercises on university sport's students so that we can have best treatment option for duration will be for 6 months, purposive sampling data will be done, subject following eligibility criteria from University of Lahore athlete students , were randomly allocated in two groups via lottery method, baseline assessment will be done, Group A participants were given baseline treatment along with foam rolling effects , Group B participants were given baseline treatment along with stretching exercises, pre or post intervention assessment will done via goniometer and Lower extremity functional scale (LESF)and three sessions per week will be given, data will be analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
The aim of the current study is to determine the effects of foam rolling versus stretching exercises on quadriceps, hamstrings and muscle length in university sport's students. It will be a Randomized control trial and will be conducted at University of Lahore. Purposive sampling technique will be used to collect data as per inclusion criteria the participant age between 18 to 25 years and male and female healthy participants. A history of cardiovascular or respiratory disease, any history of fractures or surgeries in the lower extremity in the past years will be excluded.

Patients will be randomly allocated into two groups; Group A will be treated with the effects of foam rolling on quadriceps, hamstrings and calf muscles. 5 min cycle ergometry, 6 min foam rolling 3 times for 30sec. Group B will be treated with the effects of stretching exercise on quadriceps, hamstrings and calf muscles. 5 min cycle ergometry, 6 min stretching exercises 3 times for 30sec for three sessions of treatment per week will be given. In both group's pre and post-test measurements of quadriceps, hamstrings and calf muscle length will be assessed through goniometer and Lower Extremity Functional Scale (LEFS) will be assessed to measure initial functions of lower limb. Evaluation will be done before session start and at the end of week. Total session will be given for at least 2 months.

ELIGIBILITY:
Inclusion Criteria:

* The age of participants between 18- 25 years.
* Both male and female young athletes will be included.
* Healthy participants involved

Exclusion Criteria:

* A history of cardiovascular or respiratory disease.
* Any history of fractures or surgeries in the lower extremity in the past year.
* Any history of third-degree sprains (e.g., anterior cruciate ligament ruptures), grade II or III muscle strain.
* Any prescribed medication

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Lower extremity functional scale (LEFS) | 8th Week
  It is a questionnaire containing 20 questions about the person's ability to perform task. The LESF can be used by clinicians as a measure of patient's initial function ongoing progress and outcome, as well as to set functional goals.
. Goniometric: | 8th Week
  It is an instrument which measures the available range of motion at a joint. To measure lower extremity muscles range of motion i.e. quadriceps, hamstrings and calf muscle length

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheatham SW, Stull KR. Comparison of a foam rolling session with active joint motion and without joint motion: A randomized controlled trial. J Bodyw Mov Ther. 2018 Jul;22(3):707-712. doi: 10.1016/j.jbmt.2018.01.011. Epub 2018 Feb 2. PMID 30100300
- [Background] Behara B, Jacobson BH. Acute Effects of Deep Tissue Foam Rolling and Dynamic Stretching on Muscular Strength, Power, and Flexibility in Division I Linemen. J Strength Cond Res. 2017 Apr;31(4):888-892. doi: 10.1519/JSC.0000000000001051. PMID 26121431
- [Background] Manoel ME, Harris-Love MO, Danoff JV, Miller TA. Acute effects of static, dynamic, and proprioceptive neuromuscular facilitation stretching on muscle power in women. J Strength Cond Res. 2008 Sep;22(5):1528-34. doi: 10.1519/JSC.0b013e31817b0433. PMID 18714235
- [Background] Su H, Chang NJ, Wu WL, Guo LY, Chu IH. Acute Effects of Foam Rolling, Static Stretching, and Dynamic Stretching During Warm-ups on Muscular Flexibility and Strength in Young Adults. J Sport Rehabil. 2017 Nov;26(6):469-477. doi: 10.1123/jsr.2016-0102. Epub 2016 Oct 13. PMID 27736289
- [Background] McMillian DJ, Moore JH, Hatler BS, Taylor DC. Dynamic vs. static-stretching warm up: the effect on power and agility performance. J Strength Cond Res. 2006 Aug;20(3):492-9. doi: 10.1519/18205.1. PMID 16937960
- [Background] Winters MV, Blake CG, Trost JS, Marcello-Brinker TB, Lowe LM, Garber MB, Wainner RS. Passive versus active stretching of hip flexor muscles in subjects with limited hip extension: a randomized clinical trial. Phys Ther. 2004 Sep;84(9):800-7. PMID 15330693
- [Background] McHugh MP, Cosgrave CH. To stretch or not to stretch: the role of stretching in injury prevention and performance. Scand J Med Sci Sports. 2010 Apr;20(2):169-81. doi: 10.1111/j.1600-0838.2009.01058.x. Epub 2009 Dec 18. PMID 20030776
- [Background] Bandy WD, Irion JM. The effect of time on static stretch on the flexibility of the hamstring muscles. Phys Ther. 1994 Sep;74(9):845-50; discussion 850-2. doi: 10.1093/ptj/74.9.845. PMID 8066111
- [Background] Behm DG, Chaouachi A. A review of the acute effects of static and dynamic stretching on performance. Eur J Appl Physiol. 2011 Nov;111(11):2633-51. doi: 10.1007/s00421-011-1879-2. Epub 2011 Mar 4. PMID 21373870
- [Background] Suchomel TJ, Nimphius S, Stone MH. The Importance of Muscular Strength in Athletic Performance. Sports Med. 2016 Oct;46(10):1419-49. doi: 10.1007/s40279-016-0486-0. PMID 26838985